INFORMATION AND RECEIPT OF THE VOLUNTEERS PROTOCOL

... / ... / 201 ...

In order to evaluate the impact of midwifery care based on the teaching method described in

the research on the success of breastfeeding women in postpartum period, Eskişehir

Osmangazi University Health Sciences Institute Midwifery Department student Öğr. See. It is

carried out by Arzu KUL UÇTU. Since the research is carried out with a questionnaire form,

it does not bear any risk.

You have the right to refuse to participate in the research. If you agree to participate in the

research, your answers to the questions will be kept confidential and will only be used for

research. Your answers are important to develop a valid and reliable measurement tool. It is

important to answer each question in the questionnaire given to you for the purpose of data

collection, sincerely and correctly for the reliability of the research and thank you for your

help.

RESPONSIBLE RESEARCHER

Lecturer. See. Arzu KUL UÇTU

A written and verbal statement was made to me about the text above. Under these circumstances, I agree to participate in this clinical trial with my own consent, without any

pressure or coercion.

voluntary

Name Surname: The researcher who made the explanations;

Name and surname:

Signature Signature

Address: Address:

Phone: Phone: